CLINICAL TRIAL: NCT05390333
Title: Measuring the Effectiveness of Self-Care Sampler for Family Care Partners in Reducing Caregiver Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Cigna (Unknown)
Responsible Party: Principal Investigator, Ellen Flaherty, Vice President Geriatric Center of Excellence, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02001401
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Stress
Keywords: Family Caregiver; Caregiver Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Care Sampler for Family Care Partners (Other): The 6-week Self-Care Sampler for Family Caregivers program was created to provide a variety of evidence-based self-care practices that improve the mental and physical health of caregivers by relieving stress. Sessions will take place once a week for 90 minutes, each starting with a centering exercise and focusing on a new form of self-care. The first 30 minutes will be used for a support group and the last 60 minutes will be for a self-care practice. Self-care practices that will be offered throughout the 6 weeks include mindfulness, mindful drawing, exercise, and health prevention and promotion.
  Interventions: Behavioral: Self-Care Sampler for Family Carer Partners

INTERVENTIONS:
Behavioral: Self-Care Sampler for Family Carer Partners — The 6-week Self-Care Sampler for Family Caregivers program was created to provide a variety of evidence-based self-care practices that improve the mental and physical health of caregivers by relieving stress. Sessions will take place once a week for 90 minutes, each starting with a centering exercise and focusing on a new form of self-care. The first 30 minutes will be used for a support group and the last 60 minutes will be for a self-care practice. Self-care practices that will be offered throughout the 6 weeks include mindfulness, mindful drawing, exercise, and health prevention and promotion.

SUMMARY:
To determine the effectiveness of the Self-care Sampler for Family Care Partners program in reducing caregiver stress over the 6-week program period. Hypothesis: Participants who attend the 6 class sessions over 6 weeks of the program will have a lower score on the Modified Caregiver Strain Index (MCSI) when compared to baseline. This will indicate a decrease in overall stress.

DETAILED DESCRIPTION:
The 6-week Self-Care Sampler for Family Caregivers program was created to provide a variety of evidence-based self-care practices that improve the mental and physical health of caregivers by relieving stress and encouraging preventive health behaviors (Acton, 2002). To determine the effectiveness of the Self-care Sampler for Family Care Partners program in reducing caregiver stress over the 6-week program period. Hypothesis: Participants who attend the 6 class sessions over 6 weeks of the program will have a lower score on the Modified Caregiver Strain Index (MCSI) when compared to baseline. This will indicate a decrease in overall stress. For each 6-week program, sessions will take place once a week for 90 minutes, each starting with a centering exercise and focusing on a new form of self-care. The program gives caregivers a space to connect with others and form social bonds that could extend outside of our sessions. We will run the 6-week Self-Care Sampler for Family Caregivers program three times (three intervention periods) in 2022.

ELIGIBILITY:
Inclusion Criteria:

* Any relative, partner, friend or neighbor who has a significant personal relationship with, and provides a broad range of assistance for, an older person or an adult with a chronic or disabling condition.

Exclusion Criteria:

* Those who cannot speak English which would prevent full participation
* Those with hearing, vision, or cognitive impairment that prevents participation over video
* Individuals who are not adults
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Stress, as measured by Modified Caregiver Strain Index change | Baseline, week 1 change Post-Intervention, week 6
  This index includes questions that measure the perception of persistent problems and feelings of decreased well-being that results from providing prolonged care. Respondents will provide one of the following responses to each of 13 questions:
  * Yes, on a regular basis (2 points)
  * Yes, sometimes (1 point)
  * No (0 points) These questions will be presented to the participants in a survey prior to the program and after the program. Scoring ranges from 26 to 0 with a higher score indicates a higher level of caregiver strain.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Flaherty, Ph. D, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Dartmouth Centers for Health and Aging, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acton GJ. Health-promoting self-care in family caregivers. West J Nurs Res. 2002 Feb;24(1):73-86. doi: 10.1177/01939450222045716. PMID 11829276
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Biddle S. Physical activity and mental health: evidence is growing. World Psychiatry. 2016 Jun;15(2):176-7. doi: 10.1002/wps.20331. No abstract available. PMID 27265709
- [Background] Iavarone A, Ziello AR, Pastore F, Fasanaro AM, Poderico C. Caregiver burden and coping strategies in caregivers of patients with Alzheimer's disease. Neuropsychiatr Dis Treat. 2014 Jul 29;10:1407-13. doi: 10.2147/NDT.S58063. eCollection 2014. PMID 25114532
- [Background] Jang SH, Lee JH, Lee HJ, Lee SY. Effects of Mindfulness-Based Art Therapy on Psychological Symptoms in Patients with Coronary Artery Disease. J Korean Med Sci. 2018 Mar 19;33(12):e88. doi: 10.3346/jkms.2018.33.e88. PMID 29542299
- [Background] Kabat-Zinn J. Indra's net at work: The mainstreaming of Dharma practice in society. The psychology of awakening: Buddhism, science, and our day-to-day lives. York Beach, ME, US: Samuel Weiser; 2000. p. 225-49.
- [Background] Lykins ELB, Baer RA. Psychological functioning in a sample of long-term practitioners of mindfulness meditation. Journal of Cognitive Psychotherapy. 2009;23(3):226-41. doi: 10.1891/0889-8391.23.3.226.
- [Background] Thornton M, Travis SS. Analysis of the reliability of the modified caregiver strain index. J Gerontol B Psychol Sci Soc Sci. 2003 Mar;58(2):S127-32. doi: 10.1093/geronb/58.2.s127. PMID 12646602